CLINICAL TRIAL: NCT00914381
Title: Behavioral Treatment for Cocaine Dependent Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Richard Schottenfeld, Yale University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 9410007875; R01DA006915 (NIH)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2009-06

CONDITIONS: Cocaine Dependence
Keywords: Community reinforcement approach; Contingency management; 12-step facilitation counseling; Cocaine dependence; Women
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CRA + CM (Active Comparator): Community Reinforcement Approach (CRA) combined with Contingency Management (CM)
  Interventions: Behavioral: Behavioral therapy
- TSF + CM (Active Comparator): Twelve-Step Facilitation (TSF) combined with Contingency Management (CM)
  Interventions: Behavioral: Behavioral therapy
- CRA + VC (Active Comparator): Community Reinforcement Approach (CRA) combined with Voucher Control (VC)
  Interventions: Behavioral: Behavioral therapy
- TSF + VC (Active Comparator): Twelve-Step Facilitation (TSF) combined with Voucher Control (VC)
  Interventions: Behavioral: Behavioral therapy

INTERVENTIONS:
Behavioral: Behavioral therapy

SUMMARY:
To compare the efficacy of Community Reinforcement Approach (CRA) and 12-Step Facilitation (TSF) counseling and of voucher based reward therapy (VBRT) and a yoked, non-contingent voucher control (VC) for the treatment of cocaine dependent pregnant women or women with young children.

DETAILED DESCRIPTION:
Subjects were randomly assigned to 1 of 4 treatment groups (CRA+VBRT, CRA+VC, TSF+VBRT, TSF+VC). VBRT voucher value increased for each successive cocaine-free urine sample obtained twice weekly during the 1st 12 weeks and was faded from the final earned value to $5 during the last 12 weeks. All subjects earned vouchers for attendance at scheduled twice weekly counseling sessions. Manual-guided CRA and TSF were provided by experienced clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women meeting DSM IV criteria for cocaine dependence
* Women meeting DSM IV criteria for cocaine dependence with custody of a young child

Exclusion Criteria:

* Opioid dependence
* Psychosis
* Severe depression
* Current treatment with any anti-depressant or anti-psychotic medication
* Medical instability
* Inability to understand or read English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 1994-12; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Cocaine abstinence | 24 weeks

SECONDARY OUTCOMES:
Reduced HIV risk behavior | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Schottenfeld, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - The APT Foundation, Inc. MRU, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut